CLINICAL TRIAL: NCT07328347
Title: A Simulation Experiment to Improve Dental Care for Patients With Head and Neck Tumors
Brief Title: Improving Dental Care for Patients With Head and Neck Tumors
Acronym: OncoDent
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Felix Marschner, Senior Physician, University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15/11/25
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Oral Health Care; Oral Health Behavior Change; Head & Neck Cancer; Dentist's Role; Dentist-Patient Relations
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, survey-based pre-post study conducted in two participant groups: patients with head and neck cancer and practicing dentists. Both groups complete an anonymous online questionnaire assessing knowledge, attitudes, experiences, and practices related to dental care in the context of head and neck cancer. After the baseline assessment, group-specific, guideline-based written educational information is provided. Participants then complete a post-assessment with identical content. The effect of the educational intervention is evaluated by comparing pre- and post-assessment responses within each participant group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients With Head and Neck Cancer/Dentists - Educational Information Intervention (Other): Patients with head and neck cancer and practicing dentists in Germany participate in an anonymous, prospective pre-post survey study.
  Interventions: Other: Educational material,

INTERVENTIONS:
Other: Educational material, — Patients with head and neck cancer and practicing dentists in Germany participate in an anonymous, prospective pre-post survey study. Both groups complete a baseline questionnaire assessing demographic characteristics as well as knowledge, attitudes, experiences, and decision-making related to dental care in the context of head and neck cancer treatment. Following the baseline assessment, participants receive group-specific, guideline-based written educational information. After reviewing the educational material, participants complete a post-intervention questionnaire with identical content. The effect of the educational intervention is evaluated by comparing pre- and post-assessment responses within each group.

SUMMARY:
This prospective survey study investigates knowledge, attitudes, experiences, and practices related to dental care in patients with head and neck cancer among affected patients and dentists. Participants complete an anonymous online questionnaire before and after receiving written, guideline-based information. The study aims to evaluate whether targeted educational materials improve knowledge and perceptions regarding dental care in the context of head and neck cancer treatment.

DETAILED DESCRIPTION:
This study is a prospective survey-based study using a pre-post design. Patients with head and neck cancer and practicing dentists are invited to participate. Patient recruitment is carried out through existing self-help networks and direct personal contact. National and regional self-help groups for head and neck cancer patients are contacted and asked to disseminate information about the study, including a study information sheet and a QR code linking to the online questionnaire, via their communication channels. Dentists receive an invitation letter containing the QR code to the online questionnaire by postal mail.

Participation in the study is voluntary and anonymous. By completing the online questionnaire, participants provide informed consent to participate. Due to the anonymous nature of data collection, withdrawal from the study is no longer possible after submission of the questionnaire. The survey is conducted in accordance with the data protection requirements of the Data Protection Officer of University Medical Center Göttingen, and participants are informed accordingly.

All participants initially complete a baseline questionnaire (pre-assessment) collecting demographic data as well as information on knowledge, behavior, attitudes, and experiences related to dental care for patients with head and neck cancer. Subsequently, a written educational intervention is provided. For patients, this consists of concise summaries of patient guidelines on oral cavity cancer, pharyngeal cancer, and supportive care. For dentists, the intervention includes concise summaries of relevant S3 clinical practice guidelines covering diagnosis, treatment, prevention, and follow-up of laryngeal cancer, oro- and hypopharyngeal cancer, oral cavity cancer, implant-based oral rehabilitation after head and neck radiotherapy, and supportive care in oncology.

The survey for each participant group (patients and dentists) is conducted as a single, continuous, and structured session. After accessing the educational intervention, participants are no longer able to modify their responses to the pre-assessment questionnaire. A second questionnaire with identical content is then completed (post-assessment). The effect of the educational intervention is evaluated by calculating the change (Δ) between pre- and post-assessment values.

The development of the educational interventions was informed by findings from a preceding qualitative interview study involving dentists, otolaryngologists, radiation oncologists, and patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with head and neck cancer whose health status allows completion of a questionnaire
* Practicing dentists in Germany registered in the OAK-Verlag address database

Exclusion Criteria:

* Lack of consent to participate
* Insufficient German language skills that prevent completion of the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Knowledge and Decision-Making Regarding Dental Care, Assessed by a Self-Administered Questionnaire (Percentage of Correct Responses) | Immediately after completion of the educational intervention (single study visit)
  Study outcomes are defined as the effects of the interventions measured using a self-administered questionnaire. Questionnaire responses are summarized as a percentage score ranging from 0% to 100%, with 100% indicating all responses answered correctly. For each research question, outcomes are calculated as the change (Δ) in percentage scores between pre-intervention (baseline) and post-intervention assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Göttingen, Göttingen, Germany